CLINICAL TRIAL: NCT01439282
Title: A Phase II, Multicenter, Single-Arm, Feasibility Study of Eribulin in Combination With Capecitabine for Adjuvant Treatment in Estrogen Receptor-Positive Early Stage Breast Cancer
Brief Title: Eribulin in Combination With Capecitabine for Adjuvant Treatment in Estrogen Receptor-Positive Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-212
Record Dates: First submitted 2011-09-19; First posted 2011-09-23 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2016-05

CONDITIONS: Estrogen Receptor Positive Tumor; Breast Cancer
Keywords: Estrogen Receptor-Positive Early Stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Capecitabine

ARMS (1):
- Eribulin + Capecitabine (Experimental)
  Interventions: Drug: eribulin mesylate; Drug: capecitabine

INTERVENTIONS:
Drug: eribulin mesylate — Cohort I & II: eribulin mesylate (E7389) 1.4 mg/m2 intravenously over 2 - 5 minutes on Day 1 and Day 8 for 4 cycles
  Other Names: BOLD; Halaven; E7389
Drug: capecitabine — Cohort 1: capecitabine 900 mg/m2 orally twice daily on Days 1 - 14 of a 21-day cycle for 4 cycles Cohort II: fixed dose of 1500 mg oral capecitabine twice daily, 7 days on then 7 days off for 4 cycles
  Other Names: Xeloda

SUMMARY:
This is a Phase 2, multicenter, single-arm, feasibility study evaluating eribulin in combination with capecitabine as an adjuvant chemotherapy regimen in approximately 65 subjects with early-stage (I-II), human epidermal growth factor receptor 2 (HER2)- normal, estrogen receptor (ER)-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged greater than or equal to 18 years and female subjects who must be postmenopausal (at least 12 months consecutive amenorrheic or have had a bilateral oophorectomy or, if they have had a hysterectomy but with ovaries intact, then females must be age 55 or older and with postmenopausal follicle-stimulating hormone [FSH] levels).
2. Subject is a candidate for chemotherapy in the adjuvant setting.

   * Adjuvant therapy must begin within 84 days of the final surgical procedure for breast cancer.
3. Histologically confirmed Stage I to II invasive breast cancer. Subjects may have more than one synchronous primary breast tumor.
4. Receptor Status:

   * HER2-normal as determined by a negative fluorescence in situ hybridization (FISH) result or 0 to 1+ by immunohistochemistry (IHC) staining result
   * ER-positive, node-negative or ER-positive Grade 1 or 2 node-positive breast cancer
5. ECOG performance status of 0 or 1
6. Adequate renal function as evidenced by serum creatinine less than or equal to 1.5 mg/dL or calculated creatinine clearance greater than or equal to 50 mL/min per the Cockcroft and Gault formula
7. Adequate bone marrow function as evidenced by ANC greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10.0 g/dL, and platelet count greater than or equal to 100 x 10^9/L
8. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limits of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN
9. Male subjects must have had a successful vasectomy (confirmed azoospermia), or their female partners must not be of childbearing potential, or male subjects must agree to use and have their female partners use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide] throughout the entire study period and for 30 days after study drug discontinuation..
10. Voluntary agreement to provide written informed consent and willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

1. Stage III and IV invasive breast cancer
2. Prior chemotherapy, radiation therapy, immunotherapy or biotherapy for current breast cancer
3. Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc) that would preclude any of the study therapy drugs
4. Subjects with a concurrently active second malignancy other than adequately treated nonmelanoma skin cancers or in situ cervical cancer
5. Subjects with pre-existing neuropathy greater than Grade 2
6. Subjects with known positive human immunodeficiency virus (HIV) status
7. Females of childbearing potential. Females will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrheic or have had a bilateral oophorectomy or, if they have had a hysterectomy but with ovaries intact, then females must be age 55 or older and with postmenopausal FSH levels).
8. Subjects with current gastrointestinal disease or other condition resulting in an inability to take or absorb oral medications
9. Subjects with known allergy or hypersensitivity to eribulin mesylate or its excipients, or to fluoropyrimidine therapy (with or without documented dihydropyrimidine dehydrogenase [DPD] deficiency)
10. A clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolongation of QT/QTc interval (time between the start of the Q wave and the end of the T wave/QT interval corrected for heart rate) (e.g., repeated demonstration of a QTc interval greater than 500 ms)
11. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Arizona Oncology Associates, PC - CASA, Tucson, Arizona
  - Cancer Centers of Florida, Orlando, Florida
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - New York Oncology Hematology, P.C., Albany, New York
  - Sciode Medical Associates, PLLC, d.b.a. Eastchester Center, The Bronx, New York
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology- Denton South, Denton, Texas
  - Texas Oncology-Fort Worth 12th Ave., Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology-Lewisville, Lewisville, Texas
  - Texas Oncology-Paris, Paris, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Evergreen Hematology and Oncology, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine: Eribulin mesylate (1.4 mg/m^2) was injected directly as an intravenous (IV) infusion over 2 to 5 minutes on Day 1 and Day 8 of the 21-day cycle for a total of 4 cycles. Alternatively, eribulin mesylate could be diluted in up to 100 mL in 0.9% sodium chloride for IV infusion over 2 to 5 minutes. Capecitabine (900 mg/m^2) was administered orally twice a day (BID) on Days 1 through 14 of a 21-day cycle for a total of 4 cycles. Capecitabine was to be taken approximately 30 minutes after breakfast and approximately 30 minutes after dinner.
- Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine: Eribulin mesylate (E7389) (1.4 mg/m^2) was injected directly as an IV infusion over 2 to 5 minutes on Day 1 and Day 8 of the 21-day cycle for a total of 4 cycles. Alternatively, eribulin mesylate could be diluted in up to 100 mL in 0.9% sodium chloride for IV infusion over 2 to 5 minutes. A fixed dose of capecitabine (1500 mg) was administered orally BID on a 7/7 schedule (7days on and 7 days off) for a total of 4 cycles. Capecitabine was to be taken approximately 30 minutes after breakfast and approximately 30 minutes after dinner.
Period: Overall Study
Arm/Group | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine
Started | 67 | 10
Completed | 59 | 9
Not Completed | 8 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least one dose of eribulin mesylate plus capecitabine.
Groups:
- Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine: Eribulin mesylate (1.4 mg/m^2) was injected directly as an IV infusion over 2 to 5 minutes on Day 1 and Day 8 of the 21-day cycle for a total of 4 cycles. Alternatively, eribulin mesylate could be diluted in up to 100 mL in 0.9% sodium chloride for IV infusion over 2 to 5 minutes. Capecitabine (900 mg/m^2) was administered orally BID on Days 1 through 14 of a 21-day cycle for a total of 4 cycles. Capecitabine was to be taken approximately 30 minutes after breakfast and approximately 30 minutes after dinner.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine | Total
Number analyzed (Participants) | 67 | 10 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 7 | 53
  >=65 years | 21 | 3 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 10 | 77
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved the Target Relative Dose Intensity (RDI) of 85%
Description: Relative Dose Intensity (RDI) is defined as the amount of drug administered over a specific time and is expressed as the fraction of that recommended for standard of care. The RDI for each participant was calculated as follows: (1) based on each participant's body surface area (BSA), a total planned dose for both eribulin (Dep) and capecitabine (Dcp) calculated for a full 4-cycle regimen; (2) actual total dose of eribulin (Dea) and capecitabine (Dca) for the full 4-cycle regimen as collected on the case report form; (3) overall RDI = (Dea/Dep + Dca/Dcp)/2. For each individual participant, the regimen was considered feasible if that participant was able to achieve an RDI of at least 85% of the 4 cycles of eribulin plus capecitabine treatment. Missing doses due to any reason was counted as zero in the RDI calculation.
Time Frame: 21-Day Cycle 1 through 21-Day Cycle 4
Population: Full analysis set included all participants who received at least one dose of eribulin mesylate plus capecitabine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine
Number analyzed (Participants) | 67 | 10
Percentage of participants | 77.6 [67.6 to 100] | 90.0 [60.6 to 99.5]
Statistical Analysis 1: Comparison: Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine; Test type: Superiority or Other; p = 0.1080, 1-sample binomial test — 1-side P value was obtained

2. Secondary Outcome: Use of Cold Cap for Alopecia
Description: Alopecia (hair loss) is a potential side effect of some chemotherapy agents. Chemotherapeutic drugs are toxic and could potentially harm the hair follicles (wear hair grows from) resulting in the hair falling out. It can occur in small patches on various parts of the body or all over the body and is usually temporary when related to cancer treatment. Cold cap therapy is one form of therapy for alopecia involving hair loss from the scalp. Wearing a cap or head covering with cold packs before, during, or after chemotherapy may help prevent hair loss as the cold narrows the blood vessels in the skin on your head which may lead to less of the drug reaching the hair follicles. Alopecia was one of the most common adverse events (AEs) related to eribulin only.
Time Frame: On the day of study drug infusion treatments during Cycles 1 through 4
Population: Safety analysis set included all participants who received at least one dose of study treatments and had at least one postbaseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine
Number analyzed (Participants) | 67 | 10
Participants
  Participants with alopecia | 52 | 9
  Participants who used a cold cap | 3 | 0
  Participants who did not use a cold cap | 49 | 9

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 through 30 days after last dose of study drugs (approximately up to 3 years)
Population: The safety analysis set was all participants who received at least 1 dose of study treatments and had at least 1 post treatment safety assessment.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine
Number analyzed (Participants) | 67 | 10
participants
  TEAE | 67 | 10
  SAE | 14 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events and Serious Adverse Events were collected, and included all Adverse Events with a start date on or after Day 1 through 30 days after last dose of study drugs. Participants were followed for about 1 year 3 months.
Description: TEAEs (any grade) of alopecia and neuropathy were followed until resolution or the start of another treatment whichever occurred first. AEs were graded on a 5-point scale according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Groups:
- Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine: Eribulin mesylate (1.4 mg/m^2) was injected directly as an IV infusion over 2 to 5 minutes on Day 1 and Day 8 of the 21-day cycle for a total of 4 cycles. Alternatively, eribulin mesylate could be diluted in up to 100 mL in 0.9% sodium chloride for IV infusion over 2 to 5 minutes. A fixed dose of capecitabine (1500 mg) was administered orally BID on a 7/7 schedule (7days on and 7 days off) for a total of 4 cycles. Capecitabine was to be taken approximately 30 minutes after breakfast and approximately 30 minutes after dinner.
Arm/Group | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine
Serious Adverse Events (participants affected / at risk) | 14/67 | 1/10
Other Adverse Events (participants affected / at risk) | 67/67 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine (N=67) | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine (N=10)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Eribulin Mesylate Plus 900 mg/m^2 Capecitabine (N=67) | Cohort 2: Eribulin Mesylate Plus 1500 mg Capecitabine (N=10)
Neutropenia (Blood and lymphatic system disorders) | 24 | 2
Anaemia (Blood and lymphatic system disorders) | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 0
Lacrimation increased (Eye disorders) | 9 | 0
Nausea (Gastrointestinal disorders) | 35 | 4
Diarrhoea (Gastrointestinal disorders) | 27 | 2
Constipation (Gastrointestinal disorders) | 23 | 2
Vomiting (Gastrointestinal disorders) | 15 | 0
Dyspepsia (Gastrointestinal disorders) | 10 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 1
Stomatitis (Gastrointestinal disorders) | 9 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Dry mouth (Gastrointestinal disorders) | 8 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 39 | 6
Oedema peripheral (General disorders) | 10 | 1
Pyrexia (General disorders) | 10 | 1
Mucosal inflammation (General disorders) | 8 | 2
Pain (General disorders) | 5 | 0
Asthenia (General disorders) | 6 | 0
Urinary tract infection (Infections and infestations) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 10 | 1
Alanine aminotransferase increased (Investigations) | 9 | 1
Blood bilirubin increased (Investigations) | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 0
Dehydration (Metabolism and nutrition disorders) | 10 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Headache (Nervous system disorders) | 19 | 4
Neuropathy peripheral (Nervous system disorders) | 16 | 3
Dysgeusia (Nervous system disorders) | 8 | 2
Dizziness (Nervous system disorders) | 5 | 2
Hypoaesthesia (Nervous system disorders) | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 12 | 0
Anxiety (Psychiatric disorders) | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 52 | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 27 | 2
Erythema (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 0
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 3 | 1
Local swelling (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Candida infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Electrocardiogram QT prolonged (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 2 | 1
Vision blurred (Eye disorders) | 2 | 0
Blepharospasm (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Gingival pain (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0
Early satiety (General disorders) | 1 | 0
Energy increased (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Suprapubic pain (General disorders) | 1 | 0
Tenderness (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Candidiasis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Localised infection (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Purulence (Infections and infestations) | 1 | 0
Purulent discharge (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0
Weight decreased (Investigations) | 3 | 0
Blood chloride decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Burning sensation (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Ageusia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 0
Stress (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulval ulceration (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 3 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 0
Thrombophlebitis superficial (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No